CLINICAL TRIAL: NCT01366677
Title: Development of a Yoga Intervention for Symptoms Related to Severe Visual Impairment
Brief Title: Yoga for Persons With Severe Visual Impairment
Acronym: RPY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Pamela Jeter, Postdoctoral Research Fellow, Johns Hopkins University
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: NA_00039032
Record Dates: First submitted 2011-06-02; First posted 2011-06-06 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2014-05

CONDITIONS: Sleep Disturbance; Stress; Anxiety; Depression; Balance Impairment
MeSH Terms: conditions — Parasomnias; Anxiety Disorders; Depression | interventions — Yoga

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Yoga Therapy (Experimental)
  Interventions: Behavioral: Yoga Intervention

INTERVENTIONS:
Behavioral: Yoga Intervention — Three yoga classes per week for 8 weeks.
  Other Names: Yoga, Ashtanga

SUMMARY:
This study aims to provide novel information on the feasibility of yoga interventions for secondary symptoms related to severe vision loss, such as sleep disturbances, negative mood states, fall risk and balance. This information will be important for determining safe, cost-effective and reliable practices for the benefits of yoga as an alternative means for improved health and well-being. A yoga intervention that is integrative and evidence-based will benefit the blind population through effective treatments and prevention of secondary symptoms as well as serve to inform rehabilitation specialists, educators, and clinicians in the future.

DETAILED DESCRIPTION:
This study aims to provide novel information on the feasibility of yoga interventions for secondary symptoms related to severe vision loss, such as sleep disturbances, negative mood states, fall risk and balance. This information will be important for determining safe, cost-effective and reliable practices for the benefits of yoga as an alternative means for improved health and well-being. A yoga intervention that is integrative and evidence-based will benefit the blind population through effective treatments and prevention of secondary symptoms as well as serve to inform rehabilitation specialists, educators, and clinicians in the future.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+
* Legal blindness (visual acuity worse than 20/200 but better than no/bare light perception, and/or visual field less than 20º, in the better eye)
* Any ocular disease diagnosis that is expected to remain relatively stable throughout a 3-6 month period
* Being healthy to the extent that participation yoga therapy would not exacerbate any existing disease conditions;
* Willingness to participate on a weekly basis for the 12-week intervention;
* Moderate to severe sleep disturbances, defined as ratings of 5 or greater on the PSQI

Exclusion Criteria:

* Significant changes to vision within the most recent 3-month period
* Inability to understand study procedures or communicate responses to visual stimuli in a consistent manner
* Clinically diagnosed or clinically significant sleep disorder (e.g., sleep apnea) or a medical or psychiatric condition (e.g., chronic pain) responsible for sleep complaints;
* Use of prescription sleep medication more than once a week for duration of the study;
* Use of other psychotropic medication;
* Current recipient of sleep disorder treatment;
* Consumption of more than 2-3 alcoholic beverages per day
* Smoking more than 10 cigarettes per day;

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Static Balance | Week 0 and Week 8.
  Measures will be assessed at baseline (Week 0) and immediately after the 8-week intervention at Week 8.

SECONDARY OUTCOMES:
Perceived Stress Scale | Week 0 and Week 8
  Measures will be assessed at baseline (Week 0) and immediately after the 8-week intervention at Week 8.
Profile of Mood States - Short Form | Week 0 and Week 8
  Measures will be assessed at baseline (Week 0) and immediately after the 8-week intervention at Week 8.
Exit Survey | Week 8
  The exist survey is administered immediately after the intervention during Week 8.
Fear of Falling Questionnaire | Week 0 and Week 8
  Measures will be assessed at baseline (Week 0) and immediately after the 8-week intervention at Week 8.

OTHER OUTCOMES:
Treatment Validation | Week 0, Week 4 and Week 8
  Three measures will be collected to assess the benefits of the AYT, compliance, fidelity of treatment and evaluate the participant's experience.
  1. The Philadelphia Mindfulness Scale (PHLMS).
  2. Practice/Homework Logs.
  3. Treatment Fidelity.
Physical Function | Week 0 and Week 8
  Body Mass Index (BMI), systemic blood pressure, and respiratory rate, the International Physical Activity Questionnaire (IPAQ) and flexibility measures.

CONTACTS AND LOCATIONS:
Overall Officials: Ava Bittner, PhD, OD, Principal Investigator — Johns Hopkins University
Locations (1):
- Lions Vision and Research Rehabilitation, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Jeter PE, Haaz Moonaz S, Bittner AK, Dagnelie G. Ashtanga-Based Yoga Therapy Increases the Sensory Contribution to Postural Stability in Visually-Impaired Persons at Risk for Falls as Measured by the Wii Balance Board: A Pilot Randomized Controlled Trial. PLoS One. 2015 Jun 24;10(6):e0129646. doi: 10.1371/journal.pone.0129646. eCollection 2015. PMID 26107256